CLINICAL TRIAL: NCT00003760
Title: A Phase II Trial of MGI 114 in Patients With Advanced Pancreatic Adenocarcinoma
Brief Title: Irofulvene in Treating Patients With Stage III or Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Texas (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066884; P30CA054174 (NIH); UTHSC-9895011082 (Other: UTHSCSA IRB); MGI-114.27.P98-03 (Other: Merck); SACI-IDD-98-18 (Other: San Antonio Cancer Institute); NCI-V99-1517 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Pancreatic Cancer
Keywords: stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irofulven

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irofulven — Patients receive 6-hydroxymethylacylfulvene (MGI 114) IV over 5 minutes on days 1-5. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for up to 1 year after therapy initiation.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irofulven in treating patients who have stage III or stage IV pancreatic cancer that cannot be surgically removed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the survival rate at 6 months of patients with stage III or IV unresectable adenocarcinoma of the pancreas treated with 6-hydroxymethylacylfulvene (MGI 114). II. Determine the objective tumor response rate, time to objective tumor response, and duration of response in these patients (if retrospective data is available, time to tumor progression while on prior gemcitabine is determined). III. Determine the clinical benefit of MGI 114 as measured by pain improvement, performance status, and weight. IV. Determine the survival rate at 3, 9, and 12 months in these patients. V. Gain additional information on the toxic effects and safety profile of this regimen.

OUTLINE: This is an open label, multicenter study. Patients receive 6-hydroxymethylacylfulvene (MGI 114) IV over 5 minutes on days 1-5. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed monthly for up to 1 year after therapy initiation.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage III or IV unresectable adenocarcinoma of the exocrine pancreas Must have been treated with 1 prior gemcitabine regimen, and have documented disease progression either during or within 6 months after completion of therapy Measurable or evaluable disease outside of previously irradiated area No islet cell tumors or lymphoma of the pancreas No significant CNS disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 12 weeks Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 2 mg/dL AST or ALT no greater than 2 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No atrial or ventricular arrhythmias requiring medication No atrial fibrillation (with or without medication) No ischemic event within past 6 months No history of congestive heart failure Other: Not pregnant or nursing Fertile patients must use effective contraception No significant psychiatric disorders No active infection No other prior malignancies within past 5 years, except: Basal or squamous cell skin cancer Carcinoma in situ of the cervix No concurrent serious systemic disorder

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy No concurrent immunotherapy Chemotherapy: At least 4 weeks since prior gemcitabine therapy and recovered No other prior chemotherapy (except fluorouracil as a radiation enhancing agent) No other concurrent chemotherapy Endocrine therapy: No prior hormonal therapy No concurrent hormonal therapy (except contraceptives, hormone replacement, or megestrol acetate) Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1998-11; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — San Antonio Cancer Institute
Locations (3):
- United States (3):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - San Antonio Cancer Institute, San Antonio, Texas